CLINICAL TRIAL: NCT01188655
Title: Observational Non-Interventional Study With Enbrel in Patients With Ankylosing Spondylitis
Brief Title: Observational Non-Interventional Study With Enbrel (Etanercept) in Patients With Ankylosing Spondylitis
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0881X1-4456; B1801095
Record Dates: First submitted 2010-08-24; First posted 2010-08-25 (Estimated); Results first posted 2011-04-26 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2011-09

CONDITIONS: Spondylitis, Ankylosing
Keywords: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Etanercept

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment Group Enbrel
  Interventions: Drug: Enbrel

INTERVENTIONS:
Drug: Enbrel — The patients will be treated in accordance with the requirements of the labeling of Enbrel® in Austria. The dosage and duration of therapy is to be determined by the physician to meet the patients' individual needs for treatment.
  To record complete dosing information, initial dose will be documented at baseline and any change will be documented with date, dose and reason at the subsequent visits.
  Other Names: etanercept

SUMMARY:
This observational study will be a documentation of the prescribing and administration practices of Enbrel® and their impact on ankylosing spondylitis patients outcome in a real life setting.

DETAILED DESCRIPTION:
The study population will be described using standard descriptive statistics for demographic, clinical, medical, characteristics, as well as for standard health-related quality of life and functional disability questionnaires .

ELIGIBILITY:
Inclusion Criteria:

* Proven diagnosis of Ankylosing Spondylitisin accordance with local guidelines
* Patients treated as an outpatient

Exclusion Criteria:

* Patients who suffer from hypersensitivity to the active substance Etanercept or to any of the excipients of Enbrel®.
* Treatment with Enbrel® should not be initiated in patients with active infections including chronic or localised infections.
* Patients with sepsis or risk of sepsis should not be treated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient cohort in this non-interventional study will reflect the kind of patients seen in routine clinical practice and will not be specifically pre-selected as it is the case in clinical studies.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2008-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881X1-4456&StudyName=Observational%20Non-Interventional%20Study%20with%20Enbrel%20in%20Patients%20with%20Ankylosing%20Spondylitis

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept: Participants were treated in accordance with the requirements of the labeling of Enbrel in Austria. The dosage and duration of therapy was to be determined by the physician to meet participant's individual needs for treatment. To record complete dosing information, initial dose was documented at baseline and any change was documented with date, dose and reason at the subsequent visits.
Period: Overall Study
Arm/Group | Etanercept
Started | 89
Completed | 76
Not Completed | 13
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 1
Not completed — Other | 11

BASELINE CHARACTERISTICS:
Arm/Group | Etanercept
Number analyzed (Participants) | 89
Age Continuous [Mean (Standard Deviation); unit: Years] | 41.6 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 57
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at baseline [Mean (Standard Deviation); unit: units on a scale] — BASDAI is a validated self assessment tool used to determine disease activity in participant with Ankylosing Spondylitis (AS). Utilizing a Visual Analog Scale (VAS) of 0-10 (0=none and 10=very severe) participant's answered 6 questions measuring discomfort, pain and fatigue. Number of participants analyzed for BASDAI (n)= 84
  units on a scale | 5.3 (1.6)
Bath Ankylosing Spondylitis Functional Index (BASFI) at baseline [Mean (Standard Deviation); unit: Units on a scale] — BASFI is a validated self assessment tool that determines the degree of functional limitation in AS. Utilizing a VAS of 0-10 (0 = easy, 10 =impossible), participants answered 10 questions assessing their ability in completing normal daily activities or physically demanding activities. Number of participants analyzed for BASFI (n)= 83
  Units on a scale | 4.7 (2.3)
Participant's Global Assessment Visual Analog Scale at baseline [Mean (Standard Deviation); unit: Units on a scale] — Measured using a 100mm Visual Analog Scale (VAS) ranging from 0=very good to 100=very bad. Number of participants analyzed for Participant's Global Assessment VAS (n)= 84
  Units on a scale | 6.7 (2.0)
Physician's Global Assessment Visual Analog Scale at baseline [Mean (Standard Deviation); unit: mm] — Physician Global Assessment of Disease Activity was measured on a 0 to 100 mm Visual Analog Scale (VAS), with 0 mm = no disease activity.
  mm | 6.6 (1.4)
Duration of morning stiffness at baseline [Mean (Standard Deviation); unit: minutes] — Duration of morning stiffness is defined as the time elapsed when participant woke up in the morning and was able to resume normal activities without stiffness in minutes. Number of participants analyzed for morning stiffness (n)= 80
  minutes | 88.3 (67.5)
Ankylosing Spondylitis Quality of Life Scale (ASQoL) at baseline [Mean (Standard Deviation); unit: Units on a scale] — ASQoL is a questionnaire consisting of 18 statements, related to mobility, self-care, usual activities, pain/discomfort and anxiety/depression, relevant to the physical and mental conditions of the participant with AS, to assess disease-specific quality of life. Score range: 0 (good)-18 (poor). Number of participants analyzed for ASQoL (n)= 77
  Units on a scale | 11.9 (3.9)
Percentage of Participants Without Enthesitis [Number; unit: Percentage of Participants] — Number of participants analyzed for Enthesitis (n)= 87
  Percentage of Participants | 57.5
Percentage of Participants Without Peripheral Arthritis [Number; unit: Percentage of Participants] — Number of participants analyzed for Peripheral Arthritis (n)= 87
  Percentage of Participants | 70.1
Occiput-to-wall distance [Mean (Standard Deviation); unit: centimeter (cm)] — Number of participants analyzed for occiput-to-wall distance (n)= 67
  centimeter (cm) | 3.8 (6.0)
Spine agility function by Schober test [Mean (Standard Deviation); unit: cm] — Schober test determines agility of lumbar spine. It measures participant's ability to flex lower back. Examiner makes mark at fifth lumbar vertebra (L5); places 1 finger 5 cm below and another 10 cm above the mark. Participant is asked to touch toes. Examiner measures increase in distance between 2 fingers. Number of participants analyzed (n)= 58.
  cm | 6.3 (5.5)
Spine agility function by Ott test [Mean (Standard Deviation); unit: cm] — The Ott index determines the agility of the thoracic spine. Number of participants analyzed for Ott test (n)= 48
  cm | 11.8 (14.3)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving BASDAI 40 Response at Week 24
Description: BASDAI is a validated self assessment tool used to determine disease activity in participant with Ankylosing Spondylitis (AS). Utilizing a Visual Analog Scale (VAS) of 0-10 (0=none and 10=very severe) participant's answered 6 questions measuring discomfort, pain and fatigue. The final BASDAI score averages the individual assessments for a final score range of 0-10. Participants who achieved a decrease of 40 percent or more from baseline to the following visits are called as responders.
Time Frame: Week 24
Population: Safety population: all participants who recieved at least one dose of study medication during the study period, n equals number of participants analyzed at the given time point
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 67
Percentage of participants | 83.6

2. Secondary Outcome: Change From Baseline in BASDAI at Week 12 and 24
Description: BASDAI is a validated self assessment tool used to determine disease activity in participant with Ankylosing Spondylitis (AS). Utilizing a Visual Analog Scale (VAS) of 0-10 (0=none and 10=very severe) participant's answered 6 questions measuring discomfort, pain and fatigue. The final BASDAI score averages the individual assessments for a final score range of 0-10.
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 67
units on a scale
  Week 12 (n= 70) | -2.8 (2.4)
  Week 24 (n= 68) | -3.5 (2.0)

3. Secondary Outcome: Change From Baseline in the BASFI at Weeks 12 and 24
Description: BASFI is a validated self assessment tool that determines the degree of functional limitation in AS. Utilizing a VAS of 0-10 (0 = easy, 10 = impossible), participants answered 10 questions assessing their ability in completing normal daily activities or physically demanding activities. The BASFI score is a mean score of the 10 questions.
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 83
Units on a scale
  Week 12 (n= 73) | -2.1 (2.1)
  Week 24 (n= 70) | -2.7 (2.1)

4. Secondary Outcome: Participant's Global Assessment Visual Analog Scale at Weeks 12 and 24
Description: Measured using a 100mm VAS ranging from 0=very good to 100=very bad.
Time Frame: Week 12 and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 84
Units on a scale
  Week 12 (n= 73) | 2.8 (2.2)
  Week 24 (n= 70) | 1.9 (2.2)

5. Secondary Outcome: Physician's Global Assessment Visual Analog Scale at Weeks 12 and 24
Description: Physician Global Assessment of Disease Activity was measured on a 0 to 100 mm VAS, with 0 mm= no disease activity.
Time Frame: Week 12 and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Etanercept
Number analyzed (Participants) | 89
mm
  Week 12 (n= 81) | 2.5 (1.6)
  Week 24 (n= 78) | 1.7 (1.3)

6. Secondary Outcome: Mean Duration of Morning Stiffness
Description: Duration of morning stiffness is defined as the time elapsed when participant woke up in the morning and was able to resume normal activities without stiffness in minutes (If none was present = 0; If morning stiffness was continuing, average of duration of stiffness over the past 3 days was reported; If stiffness persisted the entire day, 1440 minutes (24h x 60 minutes) was recorded).
Time Frame: Week 12 and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Etanercept
Number analyzed (Participants) | 80
minutes
  Week 12 (n= 54) | 34.2 (39.8)
  Week 24 (n= 45) | 30.0 (46.3)

7. Secondary Outcome: Change From Baseline in ASQoL at Week 12 and Week 24
Description: ASQoL is a questionnaire that assesses disease-specific quality of life (QoL). It consists of 18 statements that are relevant to the physical and mental conditions for a participant with AS: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each statement is answered by the participant as a 'Yes' (scored as 1) or 'No' (scored as 0). All item scores are summed to give a total score. Total score can range from 0 (good QoL) to 18 (poor QoL).
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 70
Units on a scale
  Week 12 | -6.8 (4.2)
  Week 24 | -8.3 (5.0)

8. Secondary Outcome: Percentage of Participants Without Enthesitis
Time Frame: Week 12 and Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 87
Percentage of Participants
  Week 12 (n= 81) | 86.4
  Week 24 (n= 78) | 85.9

9. Secondary Outcome: Percentage of Participants Without Peripheral Arthritis
Time Frame: Week 12 and Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 87
Percentage of Participants
  Week 12 (n= 81) | 81.5
  Week 24 (n= 78) | 85.9

10. Secondary Outcome: Mean Occiput-to-wall Distance at Week 12 and Week 24
Time Frame: Week 12 and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 67
cm
  Week 12 (n= 58) | 3.2 (5.5)
  Week 24 (n= 56) | 3.2 (5.2)

11. Secondary Outcome: Spine Agility Function by Schober Test
Description: Schober test determines agility of lumbar spine. It measures participant's ability to flex the lower back. Examiner makes a mark at fifth lumbar vertebra (L5); places 1 finger 5 cm below and another 10 cm above the mark. Participant is asked to touch the toes. Examiner measures the increase in distance between 2 fingers.
Time Frame: Week 12 and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 58
cm
  Week 12 (n= 50) | 7.6 (5.7)
  Week 24 (n= 49) | 7.7 (5.9)

12. Secondary Outcome: Spine Agility Function by Ott Test
Description: The Ott index determines the agility of the thoracic spine.
Time Frame: Week 12 and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 48
cm
  Week 12 (n= 40) | 13.6 (14.8)
  Week 24 (n= 43) | 13.3 (14.6)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Etanercept
Serious Adverse Events (participants affected / at risk) | 0/89
Other Adverse Events (participants affected / at risk) | 3/89
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etanercept (N=89)
Application site hypersensitivity (General disorders) | 1 (1)
Injection site erythema (General disorders) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.